CLINICAL TRIAL: NCT00554177
Title: Mifepristone After Trauma to Enhance Resilience
Brief Title: A Clinical Trial for Post Traumatic Stress Disorder
Acronym: MATTER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antonia New (Other)
Responsible Party: Sponsor-Investigator, Antonia New, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO# 07-0900
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: sexual; combat; PTSD; Clinical trial; Trauma; PTSD treatment; PTSD medication; Post traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Coitus; Wounds and Injuries | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Medicane (mifepristone)
  Interventions: Drug: Medicane (mifepristone)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Medicane (mifepristone) — 2 doses of 1200mg, Administered 2-3 days apart
  Arms: 1
Drug: Placebo — 2 doses of 1200mg, administered 2-3 days apart
  Arms: 2

SUMMARY:
he purpose of this study is to test whether a medication, called mifepristone (commonly known as the ³Morning-After-Pill²), can help to prevent emotional problems after someone has survived a traumatic experience. We are studying this medication for the treatment of Post-traumatic Stress disorder (PTSD.

DETAILED DESCRIPTION:
PTSD is an emotional illness that can develop in people after they have experienced a traumatic event. It involves symptoms such as poor sleep, nightmares about the trauma, unwanted daytime memories of the trauma (flashbacks), jumpiness, and trouble looking forward to things in the future. Once people develop PTSD, the symptoms tend to last a very long time.

We are testing the idea that mifepristone, which blocks the effect of the hormones progesterone and cortisol, will help treat PTSD. Progesterone is a hormone made in the bodies of both men and women and its main role is in regulating the menstrual cycle and in pregnancy. Cortisol is also a hormone made in the body of both men and women and helps the body respond to stress. Cortisol also has a role in making emotional memories more intense than other memories. We are testing whether blocking the effect of cortisol with mifepristone as you recall your trauma may be able to decrease the intensity of your traumatic memories. This medication will not completely block out your memories of the traumatic experience but may decrease how much your thoughts are drawn back to the memory of the traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Between 18 and 65 years old
* Have experienced one or more traumatic events within the last year €Examples for traumatic events include physical or sexual assault, combat, natural disasters, witnessing death or injury of another person, bereavement €Currently experiencing severe symptoms of anxiety including flashbacks and intrusive memories of the traumatic event. €Not currently pregnant or intending to become pregnant. If sexually active, participants must be using an approved form of birth control
* Medically healthy
* Not currently taking psychiatric medications

Exclusion Criteria:

* > Lifetime or current diagnosis of schizophrenia or other psychotic disorder, bipolar disorder, or current Axis I disorder (except for major depression secondary to the PTSD)
* Current evidence or history of significant unstable medical illness or organic brain impairment, including stroke, CNS tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, or renal or hepatic impairment.
* Patient who in the investigator¹s judgment pose a current suicidal or homicidal risk
* DSM-IV substance abuse or dependence within the past 90 days
* Patient has been taking psychotropic medication in the last 2 weeks (5 weeks for fluoxetine) prior to screening. Psychotropic medications in the last 2 weeks prior to screening, fluoxetine in last 5 weeks.
* Treatment with any other concomitant medication with primarily CNS activity
* Treatment with any medication that the PI considers not acceptable for this study.
* Patient regularly, or on average, drinks more than a) 28 units of alcohol per week for male patients, or b) 21 units of alcohol per week for female patients (1 unit = 1/2 pint of beer, or 1 glass of wine, or 1 measure of spirit)
* Pregnancy or lactation*
* Patient is currently receiving evidenced-based structured psychotherapy (e.g., cognitive-behavioral therapy, exposure therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical Administered PTSD Scale(CAPS) | once a week over eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonia New, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No